CLINICAL TRIAL: NCT03112616
Title: The Long-lasting Effects of Repetitive Neck Muscle Vibrations on Postural Disturbances in Standing Position and on Spatial Frame Reference in Chronic Stroke Patients
Brief Title: The Long-lasting Effects of Repetitive Neck Muscle Vibrations on Postural Disturbances in Standing Position in Chronic Stroke Patients
Acronym: VIBR-HEMI
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3049-VIBR-HEMI
Record Dates: First submitted 2016-08-09; First posted 2017-04-13 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Hemiplegia; Stroke
MeSH Terms: conditions — Hemiplegia; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Left-brain damaged chronic patients
  Interventions: Other: Vibration sessions
- Right-brain damaged chronic patients
  Interventions: Other: Vibration sessions

INTERVENTIONS:
Other: Vibration sessions — The patients will undergo a program of 10 sessions of vibrations of the neck muscle, each of 10 minutes, during a period of 15 days at the rate of one session per day.

SUMMARY:
One of the causes of disability in patients suffering from a stroke is postural imbalance. Sensory stimulation improves the postural symmetry of the subject transitorily and they are thought to have an effect on the spatial frame of reference through a sensory recalibration. Studies have shown that sensory stimulation by vibration of neck muscles have an immediate effect on static balance and when walking. The objective of this preliminary study is to test the long-lasting effects of repetitive neck muscle vibrations on postural disturbances in standing position and on spatial frame reference in chronic patients.

DETAILED DESCRIPTION:
The hypothesis of this study is that the proprioceptive repeated stimulation by vibration of neck muscles in the long term improved postural asymmetry in connection with the egocentric representation of body disorders.

The effect of vibration simultaneously on improving postural asymmetry and on improving markers of the perception of the body in space (LBA, SSA, Subjective Visual Vertical (SVV), Rod and frame) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years) under 80 years,
* Right or left unilateral supratentorial ischemic or hemorrhagic lesion
* The first symptomatic episode
* Stroke

  * older than 12 months
  * with or without hemianopsia
  * with or without visuospatial hemineglect
* Standing balance ≥ 30 sec unaided
* Percentage of weight bearing asymmetry on the hemiplegic lower limb (on a force platform)
* Written informed consent of the patient or a member of his entourage (in the case of patients with motor difficulties)

Exclusion Criteria:

* Orthopaedic, rheumatologic, neurologic, vestibular or visual disorders affecting the distribution of the centre of pressure while standing on the force platform
* Visual disorder that does not allow assessment of the spatial frame of reference test
* Difficulty with understanding protocol procedures

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
Changes from baseline Weight Bearing Asymmetry at Day 15 | Before and after the intervention program (Day 15)
  The primary evaluation criteria is the percentage of the Weight Bearing Asymmetry on the hemiparetic lower limb (WBA) calculated as the mean of 4 trys, each based on a 30 seconds duration with the two eyes open (OP) and then again with the two eyes closed. This evaluation is realized on a force platform.

SECONDARY OUTCOMES:
Haptic and visual Subjective Straight Ahead (SSA) test | 7 days and 15 days after the start of the intervention
  The effect on spatial reference frame evaluated by haptic and visual Subjective Straight Ahead (SSA) test
Subjective Visual Vertical (SVV) test | 7 days and 15 days after the start of the intervention
  The effect on spatial reference frame is evaluated by Subjective Visual Vertical (SVV) test
Evaluation of Longitudinal Body Axis (LBA) | 7 days and 15 days after the start of the intervention
  The effect on spatial reference frame is evaluated on Longitudinal Body Axis (LBA)
Rod and Frame Test | 7 days and 15 days after the start of the intervention
  The effect on spatial reference frame is evaluated by the Rod and Frame Test
Change from baseline of patients' motor skills | 1 month after the end of the program
  Assessment of motor skills with simple motor tasks
Change from baseline of patients' sensitivity | 1 month after the end of the program
  Assessment of superficial tact on the hemiplegic lower limb compared to the safe limb
Change from baseline of patients' spasticity | 1 month after the end of the program
  Assessment of spasticity with Ashworth Modified scale
Change from baseline of patients' functional capacity | 1 month after the end of the program
  Functional capacity is a composite index made of sensitivity test, motor scale and spasticity scale

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle BONAN, MD, PhD, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes - Pontchaillou Hospital, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No